CLINICAL TRIAL: NCT02558933
Title: Epigallocatechin Gallate (EGCG) as Therapeutic Tool to Improve Cognitive Performance in Foetal Alcohol Syndrome (FAS) Children
Brief Title: Epigallocatechin Gallate (EGCG) to Improve Cognitive Performance in Foetal Alcohol Syndrome (FAS) Children
Acronym: Neuro-SAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Óscar García-Algar, PhD, Fundacion Clinic per a la Recerca Biomédica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/5553
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2019-08

CONDITIONS: Fetal Alcohol Syndrome (FAS)
Keywords: Fetal Alcohol Syndrome; Prenatal exposure; Biomarkers; Oxidative stress; Epigallocatechin gallate
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders | interventions — epigallocatechin gallate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epigallocatechin gallate (EGCG) treated (Experimental): Intervention: Epigallocatechin gallate (EGCG) administered FAS children: An oral dose of 9 mg/Kg/day of EGCG will be administered during 1 year, with 6 control visits until 6 months after finishing the treatment
  Interventions: Dietary Supplement: Epigallocatechin gallate

INTERVENTIONS:
Dietary Supplement: Epigallocatechin gallate — Pre and post study, non randomized, controlled and without placebo, to evaluate the efficacy of Epigallocatechin gallate (EGCG). It is a pilot study in a cohort of 40 FAS children, between 7 ans 14 years old. An oral dose of 9 mg/Kg/day will be administered during 1 year, with 6 control visits until 6 months after finishing the treatment.

SUMMARY:
The flavonoid epigallocatechin gallate (EGCG) is a modulator of neuronal plasticity useful in other neurodevelopmental diseases. A recent study showed that EGCG is a promising tool for cognitive and health related quality of life improvement in Down's syndrome.

The objective is to determine the efficacy of EGCG as a therapeutic candidate for the improvement of cognitive performance in FAS patients.

Pre and post study, non randomized, controlled and without placebo, to evaluate the efficacy of EGCG. It is a pilot study in a cohort of 40 FAS children, between 7 ans 14 years old. An oral dose of 9 mg/Kg/day will be administered during 1 year, with three clinical assessments (at baseline, 6 months, and 12 months) during the treatment period.

DETAILED DESCRIPTION:
Background

1% of children present a prenatal alcohol exposure related disorder. Prevalence of consumption increases every year. In a previous study in Barcelona, 45.5% of ethanol positive meconiums were detected, as a biomarker of maternal consumption of alcohol during pregnancy. The most serious clinical picture including facial, mental and cognitive disorders is Foetal Alcohol Syndrome (FAS). Spain is the second country in adoptions from East Europe, where the consumption of alcohol during pregnancy is most important. The only prevention of FAS is avoiding consumption of alcohol during pregnancy and there is no treatment for its deleterious effects on neurodevelopment.

The flavonoid epigallocatechin gallate (EGCG) is a modulator of neuronal plasticity useful in other neurodevelopmental diseases. A recent study showed that EGCG is a promising tool for cognitive and health related quality of life improvement in Down's syndrome.

Objective To determine the efficacy of EGCG as a therapeutic candidate for the improvement of cognitive performance in FAS patients.

Methodology Pre and post study, non randomized, controlled and without placebo, to evaluate the efficacy of EGCG. It is a pilot study in a cohort of 40 FAS children, between 5 and 16 years old. An oral dose of 9 mg/Kg/day will be administered during 1 year, with three clinical assessments (at baseline, 6 months, and 12 months) during the treatment period.

Instrumentalization

1. Cognitive and neuropsychologic diagnostic scales of FAS
2. Determination of values of oxidative stress
3. Determination of control biomarkers of the treatment

ELIGIBILITY:
Inclusion Criteria:

1. FAS diagnosed children between 7 and 14 y.o.
2. Included in a previous cohort (ALMAR)
3. Informed consent by parents

Exclusion Criteria:

1. Refuse of parents to participate
2. Unfulfillment of inclusion criteria
3. Any condition in children preventing from FAS diagnostics tests application

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in values of cognitive and neuropsychologic diagnostic scales of FAS | 12 months (0, 6, and 12 months)

SECONDARY OUTCOMES:
Change of values of oxidative stress biomarkers | 6 months (0 and 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Garcia-Algar, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Joya X, Marchei E, Salat-Batlle J, Garcia-Algar O, Calvaresi V, Pacifici R, Pichini S. Fetal exposure to ethanol: relationship between ethyl glucuronide in maternal hair during pregnancy and ethyl glucuronide in neonatal meconium. Clin Chem Lab Med. 2016 Mar;54(3):427-35. doi: 10.1515/cclm-2015-0516. PMID 26351940
- [Background] Vall O, Salat-Batlle J, Garcia-Algar O. Alcohol consumption during pregnancy and adverse neurodevelopmental outcomes. J Epidemiol Community Health. 2015 Oct;69(10):927-9. doi: 10.1136/jech-2014-203938. Epub 2015 Apr 22. No abstract available. PMID 25903753
- [Background] Joya X, Garcia-Algar O, Salat-Batlle J, Pujades C, Vall O. Advances in the development of novel antioxidant therapies as an approach for fetal alcohol syndrome prevention. Birth Defects Res A Clin Mol Teratol. 2015 Mar;103(3):163-77. doi: 10.1002/bdra.23290. Epub 2014 Aug 18. PMID 25131946
- [Background] Garcia-Algar O, Black D, Guerri C, Pichini S. The effect of different alcohol drinking patterns in early to mid-pregnancy. BJOG. 2012 Dec;119(13):1670-1. doi: 10.1111/1471-0528.12007. No abstract available. PMID 23164116
- [Derived] Ramos-Triguero A, Astals-Vizcaino M, Navarro-Tapia E, Vieiros M, Bastons-Compta A, Martinez L, Andreu-Fernandez V, Garcia-Algar O. Cognitive and transcriptomic effects of Epigallocatechin gallate in fetal alcohol spectrum disorders. Sci Rep. 2026 Jan 2. doi: 10.1038/s41598-025-34576-1. Online ahead of print. PMID 41484421